CLINICAL TRIAL: NCT05438823
Title: The Effect of Technology Supported Education Program Based on Human Care Theory on Knowledge, Self-Efficacy, Quality of Life and Anxiety of Parents of Children With Stem Cell Transplantation
Brief Title: Technology Supported Education Program Based on Human Care Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Duygu ALTUNTAŞ, Lecturer, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Akdenizuni
Record Dates: First submitted 2022-06-26; First posted 2022-06-30 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-02

CONDITIONS: Stem Cell Transplantation; Nursing Caries
Keywords: caregiver; parent; stem cell transplantation; self-efficacy; quality of life; theory of human caring

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- İntervention group (Experimental): The sample of the study will be the parents of children who have had hematopoietic stem cell transplantation at Akdeniz University Hospital and whose discharge is planned (n=20).
  Interventions: Other: Educational Programe
- Control group (No Intervention): The control group will be the parents of children who underwent hematopoietic stem cell transplantation at Akdeniz University Hospital and are planned to be discharged (n=20). Participants in this group will receive routine care, and at the end of the study, training program will be applied.

INTERVENTIONS:
Other: Educational Programe — IBK-EBP will be administered to parents in six sessions in six days. After six days of training, the mobile application will be used by parents for 8 weeks. The frequency of use of the mobile application will be left entirely to the needs of the parents and reminders will be made through the mobile application. In addition, the video used during the face-to-face training, progressive relaxation exercise videos and motivational sentences will also be included in the mobile application.
  Arms: İntervention group

SUMMARY:
Hematopoietic stem cell transplantation is applied in the childhood age group for many reasons such as hematological malignancies, immune deficiencies, hemoglobinopathies, bone marrow failures and congenital metabolic diseases. The transplantation process, which requires a long hospitalization process, is an experience that causes anxiety for the child and the caregiver.

DETAILED DESCRIPTION:
It is known that during the home care process after discharge, parents experience anxiety because they are away from health professionals, and they need information and support in their care needs. This research has two purposes. 1; Developing a technology-supported home care education program (IBK-EBP) (supported by face-to-face education and mobile application) based on Human Theory of Care (IBK) for home care of children with hematopoietic stem cell transplantation. 2; It is to determine the effect of IBK-EBP education program on parents' knowledge, self-efficacy, anxiety level and quality of life. The study was planned in a single-center, follow-up, double-blind, randomized controlled design. The research sample was planned to be composed of 40 parents, 20 of which were interventions and 20 of which were controls. The home care training program, which will be prepared with up-to-date information in line with the literature; It includes face-to-face training sessions and ensuring the continuity of education at home with the mobile application to be developed. The content of the home care training program to be prepared in this context; regulation of the home environment, compliance with treatment, food safety, personal hygiene and care, social environment, planning of school life and progressive relaxation exercises. As part of the training program, parents will be shown a CD of progressive relaxation exercises before the training. Research data will be collected by a nurse other than the researchers, who was not involved in the study. Research data will be collected using the "Parent and Child Identification Form", "Parent's Knowledge Level of Care Assessment Form", "General Self-Efficacy Scale", "Quality of Life Scale for Caregivers of Cancer Patients" and "Spielberger State and Trait Anxiety Inventory". With a technology-supported home care education program to be developed based on the Human Care Theory it is predicted that the knowledge, self-efficacy, quality of life of the parents will increase and the level of anxiety will decrease, by ensuring the ease and continuity of access to information.

ELIGIBILITY:
Inclusion Criteria:

* Primary care parent of the child (0-18 years old) after HSCT
* Having mobile internet access
* Discharge planned

Exclusion Criteria:

* Parent's failure to attend at least 3 sessions of the training program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Knowledge | 1 year
  There are 13 questions in the questionnaire prepared in line with the literature. The questions will be answered as "strongly agree", "agree", "undecided", "disagree", "strongly disagree".
Self-Efficacy | 1 year
  Generalized Self-Efficacy Scale, developed by Schwarzer and Jarusalem (1995) and validated in Turkish by Aypay (2010), consists of 10 items in total. The response category is a 4-point scale and is scored as "Totally wrong = 1 point", "Slightly correct = 2 points", "Moderately correct = 3 points", "Totally correct = 4 points". There is no inverse item and cut-off point in the scale. The lowest 10 and the highest 40 points are taken from the scale. It is interpreted as "perceived self-efficacy increases as the scale score increases".
Quality Life | 1 year
  The Caregiver Quality of Life Index Cancer Scale (CQOLC), developed by Weitzner et al. (1999), aims to measure caregivers' quality of life, including their physical, emotional, familial and social functions. The total score of each sub-dimension and scale in the scale ranges from 0 to 140. In the scale, financial distress, discomfort sub-dimensions and some questions consist of reversed statements. The scale contains a total of 35 items.
Anxiety | 1 hyear
  It consists of 2 subscales, namely state and trait anxiety. State Anxiety Sub-Scale (STAI-S), an individual's at a certain time and under certain conditions; The Trait Anxiety Subscale (STAI-T) usually requires a description of how one feels. The inventory is answered via 4-point scales. The emotions and behaviors expressed in the items of the State Anxiety Sub-Scale are indicated by choosing one of the options "(1) Not at all, (2) A little, (3) A lot and (4) Completely" according to the severity of such experiences. Emotions and behaviors expressed in Trait Anxiety Sub-Scale items are according to their frequency levels; It is marked as (1) Almost Never, (2) Sometimes, (3) Often, and (4) Almost Always.

SECONDARY OUTCOMES:
Patient Satisfaction Evaluation Form According to Watson Improvement Processes | 1 year
  Watson is a form developed by Watson et al. (2010) to evaluate IBC-based nursing care. This satisfaction form is not a scale. The form consists of six questions in total. The first five questions are scored between 1 and 7, and are evaluated as never (1) and always (7). The sixth question is in the form of an open-ended question in which the "moments of care" in the given nursing care are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Proff.Dr., Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No